CLINICAL TRIAL: NCT02757690
Title: Validation and Verification of 3 Dimensional Laparoscopic System in Laparoscopic Distal Pancreatectomy & Splenectomy
Brief Title: Validation of 3 Dimensional Laparoscopic System in Disral Pancreatectomy and Splenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Song Cheol Kim, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2D vs 3D LDPS comparison
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Benign Neoplasm of Body of Pancreas; Benign Neoplasm of Tail of Pancreas

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-dimenasional distal pancreatectomy (Active Comparator): device: 2 dimensional laparoscopy of Olympus
  Interventions: Device: 2-dimensional distal pancreatectomy
- 3-dimenasional distal pancreatectomy (Experimental): device : 3 dimensional laparoscopy of Olympus
  Interventions: Device: 3-dimensional distal pancreatectomy

INTERVENTIONS:
Device: 3-dimensional distal pancreatectomy — 3D laparoscopy
  Other Names: 3D
  Arms: 3-dimenasional distal pancreatectomy
Device: 2-dimensional distal pancreatectomy — 2D laparoscopy
  Other Names: 2D
  Arms: 2-dimenasional distal pancreatectomy

SUMMARY:
Traditionally, laparoscopy has been based on 2-dimensional (2D) imaging, which has represented a considerable challenge for those approaching this technique. Thus, 3-dimensional (3D) visualization technology for laparoscopy has been proposed, since the early 1990s, as a way to facilitate laparoscopic performance. However, early 3D laparoscopic technology was limited in terms of image quality, so that its use had not been implemented. More recently, industry has developed novel 3D systems where the imaging is similar to stereoscopic vision, in which the depth perception is achieved by different unique images received by each eye. Thus, more recent studies have suggested a possible advantage provided by these new 3D systems during laparoscopic performance. However, comparative assessments of new generation 3D vs 2D laparoscopy remain limited, especially in the hepatobiliary and pancreatic field.

To assess the benefits and harms of use of three dimensional systems versus two dimensional systems during laparoscopic distal pancreatectomy.

DETAILED DESCRIPTION:
Procedures

1. the investigators will take the patient consent for this clinical trial.
2. The participants will be divided with two groups with block randomized method
3. Skillful pancreatic surgeon will perform 2D or 3D laparoscopic distal pancreatectomy.
4. The participants will be monitor the intraoperative and postoperative course.

Data collection

1. operation video : operation time, number of errors (missed grasp, loss of material)

   1. Segmental operation time according to procedure
   2. Numbers of errors during operation
2. clinical parameters:

   1. Blood examination : complete blood count (hemoglobin, white blood cell count), amylase, lipase, etc.
   2. Radiological examination: X-ray, Computed Tomography (CT), Magnetic Resonance Imaging (MRI), etc
   3. Medical records : hospital stay after operation, the time to eating, pathologic examination
3. Subjective scoring in the view of operator, 1st assist.

   1. Scoring for imaging quality
   2. Scoring for harms of 3D/2D laparoscopic system
   3. Scoring for overall demand

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 (Kg/m2)
* History of severe or recurrent pancreatitis
* Mass size > 10cm
* History of low abdomen major operation
* Additional resection for extra-pancreatic organ

Exclusion Criteria:

* Participants refusal.
* Additional resection dependent on pathological examination in intraoperative or postoperative period.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Operation time | expected duration: 200mins (for each operation)
  The unedited videos of the operations will be assessed from start to end of the operation by two clinicians. The average of operation time will be compare according to 2D versus 3D laparoscopic system.

SECONDARY OUTCOMES:
Numbers of errors during operation | During operation (expected duration: 200mins)
  The investigators will check the error number of operator during operation with review the video record of the operation
Subjective scoring in the view of operator, 1st assist | During operation (expected duration: 200mins)
  The investigators will check the subjective scoring of operator and 1st assist during operation. For example, depth perception, sharpness, visual strain, headache, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Songcheol Kim, MD PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: Undecided